CLINICAL TRIAL: NCT01889823
Title: Effects of Oxygen Status on Hypoxia Inducible Factor 1-α and Inflammation. A Pilot Proof of Principle Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Peter Pickkers, Prof. dr. P. Pickkers, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OX1
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Hypoxia; Hyperoxia
Keywords: Oxygen; Hypoxia; Hyperoxia; Inflammation; Innate immunity
MeSH Terms: conditions — Hypoxia; Hyperoxia; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypoxia (Experimental): Subjects will be breathing an individualized mix of nitrogen and room air titrated to an oxygen saturation of 80-85%.
  Interventions: Other: Hypoxia
- Hyperoxia (Experimental): Subjects will be breathing 100% of oxygen
  Interventions: Other: Hyperoxia

INTERVENTIONS:
Other: Hypoxia — Subjects will be breathing an individualized mix of nitrogen and room air titrated to an oxygen saturation of 80-85%.
  Arms: Hypoxia
Other: Hyperoxia — Subjects will be breathing 100% oxygen
  Arms: Hyperoxia

SUMMARY:
It has been shown in in vitro and animal models that hypoxia can have pro-inflammatory effects and hyperoxia can have anti-inflammatory effects. The pro-inflammatory effect could be the result of activation of Hypoxia Inducible Factor, a transcription factor that is known to activate many cell systems aimed at cell survival, including the inflammatory response. The anti-inflammatory effects of hyperoxia could be the annihilation of Hypoxia Inducible Factor, but also a decrease in inflammation due to oxygen toxicity resulting in a decrease in clearance of pathogens. These effects have been sparsely studied in humans. Therefore, we hypothesize that hypoxia results in an increase in Hypoxia Inducible Factor in circulating leukocytes and increases inflammatory reactions, whereas hyperoxia decreases these reactions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤35 yrs
* Male
* Healthy

Exclusion Criteria:

* Use of any medication
* Smoking
* History, signs or symptoms of cardiovascular disease
* History of atrial or ventricular arrhythmia
* (Family) history of myocardial infarction or stroke under the age of 65 years
* Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrioventricular block or a complex bundle branch block
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90 mmHg)
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50 mmHg)
* Renal impairment (defined as plasma creatinine >120 μmol/l)
* Liver enzyme abnormalities alkaline phosphatase>230 U/L and/or ALT>90 U/L
* Medical history of any obvious disease associated with immune deficiency
* CRP > 20 mg/L, WBC > 12x109/L, or clinically significant acute illness, including infections, within 4 weeks before endotoxemia day
* Participation in a drug trial or donation of blood 3 months prior to the experiment
* Pre-existent lung disease or asthma
* Use of recreational drugs within 21 days prior to experiment day
* Visit to altitude >1500m within 4 weeks prior to the experiment
* Air travel with flight time over 3 hours within 4 weeks prior to the experiment
* History of acute mountain sickness
* Recent hospital admission or surgery with general anaesthesia (<3 months)
* Claustrophobia
* Feelings of discomfort during a 10 minute test wearing the transparent respiratory helmet at the screening visit

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Hypoxia Inducible Factor 1 alpha in circulating leukocytes | 24 hours
  Hypoxia Inducible Factor 1 alpha in circulating neutrophils, lymphocytes and monocytes as measured with flow cytometry

SECONDARY OUTCOMES:
Hypoxia Inducible Factor mRNA and anti Hypoxia Inducible Factor mRNA in circulating leukocytes | 24 hours
Reactive Oxygen Species in circulating leukocytes | 24 hours
  ROS in circulating leukocytes, subclassified in neutrophils and monocytes
Phagocytic function of circulating leukocytes | 24 hours
cytokine production after ex vivo stimulation of leukocytes | 24 hours
circulating cytokines (including but not limited to IL-6, IL-10, IL-1RA) | 24 hours
Hemodynamic parameters | 24 hours
  Blood pressure, heart frequency, cardiac output measurement
ventilatory response | 24 hours
  Measures of ventilation: respiratory rate, blood gas changes
adenosine metabolism | 24 hours
  urine and plasma adenosine,adenosine receptor mRNA, purines
alkaline phosphatase | 24 hours
cognitive function | 24 hours
  neuropsychologic assessment of cognitive function
Hepcidin and iron parameters | 24 hours
catecholamines | 24 hours
  adrenaline, noradrenaline and dopamine
Neutrophil function | 24 hours
body temperature | 24 hours
oxygen saturation and PaO2 | 24 hours
subjective symptoms | 24 hours
high sensitive troponin | 24 hours
iFABP | 24 hours
Brain specific proteins | 24 hours
endocan | 24 hours
adrenomedullin | 24 hours
EPO | 24 hours
VEGF | 24 hours
Heart rate variability | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dorien Kiers, MD, Principal Investigator — Intensive Care Medicine, Radboud University Nijmegen Medical Centre; Peter Pickkers, MD,PhD, Study Director — Intensive Care Medicine, Radboud University Nijmegen Medical Centre
Locations (1):
- Intensive Care Medicine, Radboud University Nijmegen Medical Centre, Nijmegen, Nijmegen, Gelderland, Netherlands